CLINICAL TRIAL: NCT05972967
Title: A Phase 2 Proof of Concept Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of OMS906 in PNH Patients With a Sub-optimal Response to the C5 Inhibitor, Ravulizumab
Brief Title: Safety and Efficacy of OMS906 in Paroxysmal Nocturnal Hemoglobinuria Patients With a Sub-optimal Response to Ravulizumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Omeros Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OMS906-PNH-001
Record Dates: First submitted 2023-07-11; First posted 2023-08-02 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: PNH
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 3 mg/kg IV OMS906 with Ravulizumab IV (Experimental): Up to 6 doses of 3 mg/kg at 8-week intervals. All patients will receive 3 doses of OMS906 of 3 mg/kg Intravenous (IV) at 8-week intervals. Clinical responders at Week 24 will receive an additional 3 doses of OMS906 only at 8-week intervals at 5 mg/kg (monotherapy). Incomplete responders may receive an additional 3 doses of OMS906 with ravulizumab at 8-week intervals. Non responders will not receive additional OMS906.
  Interventions: Biological: OMS906
- 5 mg/kg IV OMS906 with Ravulizumab IV (Experimental): Up to 6 doses of 5 mg/kg at 8-week intervals. All patients will receive 3 doses of OMS906 of 5 mg/kg Intravenous (IV) at 8-week intervals. Clinical responders at Week 24 will receive an additional 3 doses of OMS906 only at 8-week intervals (monotherapy). Incomplete responders may receive an additional 3 doses of OMS906 with ravulizumab at 8-week intervals. Non responders will not receive additional OMS906.
  Interventions: Biological: OMS906

INTERVENTIONS:
Biological: OMS906 — Biological: OMS906
  Other Names: zaltenibart

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics, pharmacodynamics and preliminary efficacy of OMS906 for the treatment of Paroxysmal Nocturnal Hemoglobinuria (PNH) in patients who have a sub-optimal response to ravulizumab.

DETAILED DESCRIPTION:
This is a Phase 2, proof of concept, open label study examining two doses of OMS906, 3 mg/kg and 5 mg/kg IV given to PNH patients at 8-week intervals, first in combination with the C5 inhibitor ravulizumab then as monotherapy. The primary objective is to assess overall safety and tolerability of repeat-dose IV OMS906 administration at 8-week intervals in patients with PNH.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of PNH by flow cytometry with PNH clone size of > 10% red blood cells (RBCs) and/or granulocytes.
2. Male or female adults 18 years and older.
3. Completed informed consent procedures.
4. In relation to ravulizumab treatment prescribed in accordance with its marketing authorization and summary of product characteristics (SmPC):

   • Must have a sub-optimal response to ravulizumab, defined as a hemoglobin level < 10.5 g/dL despite treatment measured at screening and confirmed at baseline (Day 1, predose). Ravulizumab treatment will have been maintained at a stable dose for at least 2 doses (4 months) prior to baseline.
5. Female patients of child-bearing potential must have a negative highly sensitive urine pregnancy test at screening and prior to each dose of OMS906.
6. Females must use highly effective birth control to prevent pregnancy during the clinical trial and for 20 weeks (140 days) following their last dose of study drug. If a female, must be sterile (either surgically or biologically)* or at least one year postmenopausal**, or have a monogamous partner who is surgically sterile, or have a same sex partner, or if in a heterosexual relationship, must agree to comply with the following contraception guidelines:

   * Practice abstinence (only considered an acceptable method of contraception when it is in line with the patients' usual and preferred lifestyle and the patient agrees to refrain from heterosexual intercourse during the entire period of risk associated with the study treatments, including during the clinical trial and for 20 weeks [140 days] following their last dose of study drug), or
   * Use at least 1 of the following medically acceptable methods of birth control:

     * Hormonal methods as follows:

   Combined estrogen and progestogen containing hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal). Progestogen only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
   * Intrauterine devices
   * Intrauterine hormone-releasing systems
   * Vasectomized partner * Defined as having had a hysterectomy and/or bilateral oophorectomy, bilateral salpingectomy or bilateral tubal ligation/occlusion at least 6 weeks prior to screening; or have a congenital or acquired condition that prevents childbearing.

     * Defined as at least 12 months with no menses without an alternative medical cause) [can be confirmed with follicle stimulating hormone level (FSH) in the postmenopausal range (FSH levels ≥40 milli-International unit (mIU)/mL at Screening) if the patient is not using hormonal contraception or on hormonal replacement therapy]. In the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.
7. Males must use highly effective birth control with a female partner to prevent pregnancy during the clinical trial and for 20 weeks (140 days) following their last dose of study drug that include the following:

   * Practice abstinence (only considered an acceptable method of contraception when it is in line with the patients' usual and preferred lifestyle and the patient agrees to refrain from heterosexual intercourse during the entire period of risk associated with the study treatments, including during the clinical trial and for 20 weeks [140 days] following their last dose of study drug), or
   * Use (or have their partner use) acceptable, highly effective contraception (see Criterion #6) during heterosexual activity.

Exclusion Criteria:

1. History of major organ transplant or hematopoietic stem cell/marrow transplant.
2. Platelet count < 30,000/µL or absolute neutrophil count < 500 cells/µL at Screening.
3. Anemia, as evidenced by hemoglobin < 10.5 g/dL, attributable to any other medical condition apart from PNH.
4. Elevation of liver function tests, defined as total bilirubin > 2×ULN, direct bilirubin > 1.5× upper limit of normal (ULN), and elevated transaminases, alanine aminotransferase (ALT) or aspartate aminotransferase (AST), > 2×ULN unless due to PNH related hemolysis.
5. History of any severe hypersensitivity reactions to other monoclonal antibodies or excipients included in the OMS906 preparation.
6. Significant active bacterial or viral infection within the 2 weeks prior to Screening, including COVID-19 infection.
7. Immunodeficiency or immunosuppression (including chronic use of immunosuppressive drugs, such as ciclosporin or tacrolimus).
8. History of meningococcal disease and/or has not received vaccination for N. meningitidis.
9. Pregnant, planning to become pregnant, or nursing female patients.
10. Recent surgery requiring general anesthesia within the 2 weeks prior to Screening or expected to have surgery requiring general anesthesia during the Treatment Period.
11. History of any significant medical, neurologic, or psychiatric disorder that in the opinion of the Investigator would make the patient unsuitable for participation in the study.
12. Treatment with any investigational medicinal product or investigational device within 30 days (or within 5× its half-life in days, whichever is the longer period) prior to Screening, or participation in another concurrent clinical trial involving a therapeutic intervention. Participation in observational and/or registry studies is permitted.
13. Unable or unwilling to comply with the requirements of the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
To assess the overall OMS906 administration at 8-week intervals in PNH patients. | 56 weeks
  Number and % of participants with Treatment-emergent Adverse Events (TEAEs) as assessed by CTCAE v5.0, including abnormalities in laboratory measures, ECGs and physical examinations

SECONDARY OUTCOMES:
Incidence of patients with hemoglobin increase ≥ 2.0 g/dL from baseline (Response criterion) baseline on adjunctive treatment and sustained during monotherapy. | 56 weeks
  Number and % of participants with hemoglobin increase ≥ 2.0 g/dL from baseline on adjunctive treatment and sustained during monotherapy
Reticulocyte count | 56 weeks
  Individual patient changes from baseline in absolute reticulocyte counts
Lactate dehydrogenase (LDH) | 56 weeks
  Individual patient changes from baseline in LDH
Transfusion requirements | 56 weeks
  Number of transfusions required during each treatment phase will be compared with the transfusion history prior to the study
Pharmacokinetics (PK) of multiple-dose administration of OMS906 | 56 weeks
  PK parameters including OMS906 maximum concentration (Cmax) and Area under the plasma concentration versus time curve (AUC)
Pharmacodynamics (PD) of multiple-dose administration of OMS906 | 56 weeks
  Mature Complement Factor D (CFD) concentration
OMS906 anti-drug antibodies (ADA) | 56 weeks
  Number of patients with measurable ADA

CONTACTS AND LOCATIONS:
Overall Officials: Edward Philpot, MD, Study Director — Omeros Corporation
Locations (5):
- Germany (2):
  - Omeros Investigational Site, Aachen
  - Omeros Investigational Site, Ulm
- Omeros Investigational Site, Thessaloniki, Greece
- Omeros Investigational Site, Lausanne, Switzerland
- Omeros Investigational Site, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No